CLINICAL TRIAL: NCT04985227
Title: Impact of Home Weight Tele-monitoring on the Number of Office Visits in the First Six
Brief Title: Impact of Home Weight Tele-monitoring on the Number of Office Visits in the First Six Weeks of Life in Infants.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: American Academy of Pediatrics (Other)
Responsible Party: Principal Investigator, Anirudha Das, Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21-583
Record Dates: First submitted 2021-07-23; First posted 2021-08-02 (Actual); Last update posted 2023-03-13 (Actual); Status verified 2023-03

CONDITIONS: Failure to Thrive; Newborn Morbidity
MeSH Terms: conditions — Failure to Thrive

STUDY DESIGN:
Intervention Model Description: Randomized controlled Trial. One group has no intervention. Second group will be provided with a weighing scale and ask to report the infant's weight back to the provider.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home weight monitoring (Experimental): Weighing scales will be provided to the parents to weigh their infant and enter the weight daily during the weekdays into the patient portal.
  Interventions: Other: Home weight monitoring
- Control (No Intervention): The parents will visit their Primary Care office in the usual manner as recommended by their Pediatrician.

INTERVENTIONS:
Other: Home weight monitoring — Parents will be provided with weighing scales to weigh their infant at home and plug in the weight in the patient portal for review by their primary care provider.
  Arms: Home weight monitoring

SUMMARY:
Currently American Academy of Pediatrics (AAP) Bright Futures Guideline recommends 2 visits for all healthy term newborn infants in the first 6 weeks of life, first at 3-5 days of life and the second at around a month. However, compliant parents of infants are known to get at least 1-2 extra visits due to primary care provider's concern about appropriate weight gain. These weight check visits as they take up extra time, car gas, parking charges, loss of work time and paying for childcare during the visits. Clinic resources are also unnecessarily utilized. Remote home monitoring of infant weights with the use of technology could reduce the need for office visits and improve efficiency on the provider side, enhance parental satisfaction and decrease transmission of viruses in the winter season. The main objective is to monitor the daily weight of term infants born at 37 completed weeks of greater, discharged from the newborn nursery, remotely through the electronic medical record by the primary care provider and to reduce any extra visit in the first six weeks of life. Using block randomization, the infants will be assigned to either group A, where no home telemonitoring of weight will take place or group B, where the parent will be provided with a weighing scale. The parent will enter the weight into the MyChart application on the smartphone or on the computer which will be tracked by the pediatrician. The pediatrician will take the decision whether to bring the infant in for a weight check visit based on the weight information. If the weight gain is satisfactory, the pediatrician will see the patient at around 1 month of age per recommendation and the parents will stop the weight checks at that time. The sample size required was 16 on each arm (total 32) which has been increased to 20 each arm to account for technical problems and/or loss to follow up.

DETAILED DESCRIPTION:
Title: Impact of a pilot home weight telemonitoring program on the number of office visits by infants in the first six weeks of life

Purpose: Currently American Academy of Pediatrics (AAP)Bright Futures Guideline recommends five health supervision or office visits in the first 6 months of life for infants discharged from the newborn nursery. This includes 2 visits in the first 6 weeks, first at 3-5 days of life and the second at around a month.1 However, compliant parents of infants are known to get at least 1-2 extra visits due to primary care provider's concern about appropriate weight gain. These weight check visits are an inconvenience to the parent(s) as they not only take up extra time, but also utilize the limited resources these parents have. Travel car gas, parking charges, loss of work time and paying for childcare during the visits are some of the ways the finances are affected. There is also utilization of resources in the clinic, as well as time slots that could be utilized to see other patients. Previous studies have shown greater maternal satisfaction with effective telemonitoring of weight at home.2,3 Remote home monitoring of infant weights with the use of technology could reduce the need for office visits and improve efficiency on the provider side, enhance parental satisfaction and decrease transmission of viruses in the winter season. Reduction in the number of visits to the outpatient visit may also help in curbing the spread of coronavirus in the pandemic.

Objectives:

1. To monitor the daily weight of infants remotely through the electronic medical record by the primary care provider.
2. To reduce any extra visit in the first six weeks of life of an infant other than those recommended by AAP, primarily for a concern of appropriate weight gain.

Target population: Newborns with gestation of 37 weeks and zero days or more, discharged from the newborn nursery who will follow-up with a clinician within the Cleveland Clinic health system (CCHS).

Proposal: Institutional Review Board approval will be obtained before the study initiation. The study will require taking consent from parent.

Methods: In a prospective pilot randomized controlled study, using computer generated randomization, infants born at Fairview Hospital meeting the inclusion criteria will be randomized to either group A (home telemonitoring of daily weight, scale provided to parents) or group B (no home telemonitoring, no scale provided). If the infant falls in the group A, the parent(s) of the infant will be given a weighing scale before discharge from the newborn nursery at Fairview Hospital with detailed instructions on how to use the scale. The instructions will be in English only. The parent(s) will be requested to document daily weight (at least 5 days a week) till the 1 month visit of the infant to the Pediatrician.

Study population/workflow process:

The parent(s) in group A will be provided with the instructions on how to weigh their infant and document the weight in patient portal provided by the Cleveland Clinic. The entire process will be demonstrated to the parent(s) in the newborn nursery prior to discharge. The daily weight will be monitored by the pediatrician via the flowsheet through the electronic medical record (EMR). The infant's pediatrician is defined as the first clinician (Physician or Nurse Practitioner) the infant visits at the outpatient visit after discharge from the newborn nursery.

The parent could also call the office with concerns about weight gain as instructed by the pediatrician's office. If the weight gain of the infant is appropriate, the pediatrician will continue to monitor and see the infant at 1 month of life as recommended by the AAP. But if there are any concerns, the provider will be free to intervene as per his/her discretion. The parent will stop weight documentation after the 1-month pediatrician visit. The number of visits needed by infants will be compared between the groups at the 6 months mark.

Data and safety monitoring plans:

The research study entails use of a standard commercially available weighing scale for use at home by the parent. If used correctly, this intervention poses less than minimal risk to the infant. All the communication that will take place between the provider and the parent will be through HIPAA compliant platforms - MyChart and Epic. Parents' will be encouraged to contact the PI directly for any concerns about the process of weighing or safety of the data. All data will be stored in HIPAA compliant RedCap database.

Informed consent:

An IRB approved consent form in English will be used. The consent interview will take place in the parents' private room in the Fairview 4 North unit. Sufficient time will be provided to the parent to make a decision about participating in the study. The consent interview will be conducted by the study PI or the co-investigator. The consent will be documented in an IRB approved consent document.

The parent of the subject (newborn) will be provided with information regarding the research. If the treating team allows the mother to take her baby home with her, it will be assumed that the mother is the responsible guardian who is able to give consent for the study. The capacity to consent will be decision that will be made by the study team after consultation with the treating team of the mother and baby.

Risks benefits:

There is a risk of breach in confidentiality because of the data leak from being transmitted from the smartphone MyChart app to the electronic medical record. The use of the MyChart app is guided by the standard agreements/terms of use/privacy policy of the Cleveland clinic. All standard precautions including compliance to HIPAA will apply to this process of data transfer. Therefore, the research does not involve no more than the standard security risks that apply to the use of MyChart application.

The information will be kept confidentially in a HIPAA compliant data repository, RedCap. After the study is completed, the data will be destroyed or de-identified. All data will be coded before analysis. Any personal information that could identify individuals will be removed or changed before files are shared with other researchers or results are made public.

Participation in this study may or may not benefit the infant directly by reducing the number of times the infant would have to visit the Pediatrician in-person, depending on his/her study group. But participation in this study may provide information that may reduce the number of visits required for infants to visit their doctors in-person in the first month of life. The knowledge to be gained from this research may be beneficial for other patients.

Costs:

There are no charges to be billed for the research. The only cost of the study is the purchase of 20 weighing scales for which adequate funding is available. The PI and Co-investigators will manage to take consent and follow the 20 infants who will be in group A (weighed by the scale). Statistical analysis will be performed by the PI. No other cost is expected in the study.

Statistical analysis: The aim is to demonstrate a difference of 1 visit in the first 6 weeks of life between the groups (2 vs 3). Considering an alpha of 0.05 and a power of 80%, 16 infants in each group [16 with weighing scales (group A) and the 16 without (Group B)] will be needed. Considering 25% loss of follow-up due to technical issues or drop-out, our total subjects is estimated to be 20 subjects in each group (total 40). The parents will be instructed to document 5 weight measurements in a week but an Intent to treat analysis will be utilized to include all infants in Group B who have weight documentation < 5 times in a week.

Funding: The study is funded by AAP district V SONPM grant program.

ELIGIBILITY:
Inclusion Criteria:

1. Born at Fairview Hospital and discharged from the newborn nursery
2. Gestation of 37 weeks and 0 days or greater and weight appropriate for gestation age
3. Weight loss is within the range of normal per standard guidelines for the postnatal day (need to elaborate)
4. Parents who agree to download the patient portal application of Cleveland Clinic and have access to the infant's information on it.

Exclusion Criteria:

1. Admitted to the NICU after birth
2. Congenital malformations or complex health care issues requiring outpatient monitoring by any other provider other than the pediatrician.
3. History of drug abuse in mother
4. Twin or triplet birth
5. Mother does not speak English

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-02-24 (Actual)

PRIMARY OUTCOMES:
Number of visits | 1 month
  Number of visits to the Primary Care providers office in the first month of life

CONTACTS AND LOCATIONS:
Overall Officials: Anirudha Das, Principal Investigator — The Cleveland Clinic
Locations (1):
- Fairview Hospital, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data will be stored in a data repository and shared with the journal

REFERENCES:
- [Background] DiTomasso D, Roberts M, Parker Cotton B. Postpartum Mothers' Experiences With Newborn Weight Checks in the Home. J Perinat Neonatal Nurs. 2018 Oct/Dec;32(4):333-340. doi: 10.1097/JPN.0000000000000367. PMID 30216202
- [Background] DiTomasso D, Ferszt G. Mothers' Thoughts and Feelings About Using a Pediatric Scale in the Home to Monitor Weight Changes in Breastfed Newborns. Nurs Womens Health. 2018 Dec;22(6):463-470. doi: 10.1016/j.nwh.2018.10.004. Epub 2018 Oct 30. PMID 30389281
- See also: AAP Bright futures periodicity schedule — https://www.aap.org/en-us/professional-resources/practice-transformation/managing-patients/Pages/Periodicity-Schedule.aspx